CLINICAL TRIAL: NCT03323034
Title: A Phase 1 Study of Pevonedistat (MLN4924), a NEDD8 Activating Enzyme (NAE) Inhibitor, in Combination With Temozolomide and Irinotecan in Pediatric Patients With Recurrent or Refractory Solid Tumors
Brief Title: Pevonedistat, Irinotecan, and Temozolomide in Treating Patients With Recurrent or Refractory Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL1615; NCI-2017-01229 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ADVL1615; ADVL1615 (Other: Pediatric Early Phase Clinical Trial Network); ADVL1615 (Other: CTEP); UM1CA097452 (NIH)
Record Dates: First submitted 2017-10-11; First posted 2017-10-26 (Actual); Results first posted 2022-09-23 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Recurrent Lymphoma; Recurrent Malignant Solid Neoplasm; Recurrent Primary Central Nervous System Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Primary Central Nervous System Neoplasm
MeSH Terms: conditions — Lymphoma; Central Nervous System Neoplasms | interventions — Irinotecan; pevonedistat; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pevonedistat, temozolomide, irinotecan) (Experimental): Patients receive pevonedistat IV over 60 minutes on days 1, 8, 10, and 12, temozolomide PO daily on days 8-12, and irinotecan IV over 90 minutes on days 8-12 of cycle 1. Beginning cycle 2, patients receive pevonedistat IV over 60 minutes on days 1, 3, and 5, temozolomide PO daily on days 1-5, and irinotecan IV over 90 minutes on days 1-5. Treatment repeats every 28 days for cycle 1 and 21 days for subsequent cycles for up to 17 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Irinotecan; Drug: Pevonedistat; Drug: Temozolomide

INTERVENTIONS:
Drug: Irinotecan — Given IV
Drug: Pevonedistat — Given IV
  Other Names: MLN4924; Nedd8-Activating Enzyme Inhibitor MLN4924
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase I trial studies the side effects and best dose of pevonedistat when given together with irinotecan hydrochloride and temozolomide in treating patients with solid tumors, central nervous system (CNS) tumors, or lymphoma that have come back after a period of improvement (recurrent) or that do not respond to treatment (refractory). Pevonedistat and irinotecan may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pevonedistat, irinotecan hydrochloride, and temozolomide may work better in treating patients with solid tumors, central nervous system (CNS) tumors, or lymphoma compared to irinotecan and temozolomide alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of pevonedistat administered as an intravenous infusion on days 1, 8, 10, and 12 of a 28-day cycle (cycle 1), and on days 1, 3, and 5 of a 21-day cycle (cycle 2 and beyond) in combination with irinotecan (administered as an intravenous infusion on days 8-12 of cycle 1 and days 1-5 of cycles 2+) and temozolomide (administered orally on days 8-12 in cycle 1 and days 1-5 of cycles 2+) in children with recurrent or refractory solid tumors, including central nervous system (CNS) tumors and lymphoma.

II. To define and describe the toxicities of pevonedistat administered on this schedule.

III. To characterize the pharmacokinetics of pevonedistat in children with recurrent or refractory cancer.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of pevonedistat within the confines of a phase 1 study.

II. To assess the biologic activity of pevonedistat.

OUTLINE: This is a dose escalation study of pevonedistat.

Patients receive pevonedistat intravenously (IV) over 60 minutes on days 1, 8, 10, and 12, temozolomide orally (PO) daily on days 8-12, and irinotecan IV over 90 minutes on days 8-12 of cycle 1. Beginning cycle 2, patients receive pevonedistat IV over 60 minutes on days 1, 3, and 5, temozolomide PO daily on days 1-5, and irinotecan IV over 90 minutes on days 1-5. Treatment repeats every 28 days for cycle 1 and 21 days for subsequent cycles for up to 17 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Part A1: Patients must be >= 12 months and =< 21 years of age at the time of study enrollment
* Part A2: Patients must be >= 6 months and < 12 months of age at the time of study enrollment; patients will enroll one dose level behind the dose level at which patients in Part A1 are enrolling
* Patients with recurrent or refractory solid tumors, including CNS tumors and lymphoma, for which no standard therapy is available are eligible; patients must have had histologic verification of malignancy at original diagnosis or relapse except in patients with intrinsic brain stem tumors, optic pathway gliomas, or patients with pineal tumors and elevations of cerebrospinal fluid (CSF) or serum tumor markers including alpha-fetoprotein or beta-human chorionic gonadotropin (HCG)
* Patients must have either measurable or evaluable disease
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; NOTE: neurologic deficits in patients with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment; if after the required time frame, the numerical eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive; at least 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea); the duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil counts [ANC] counts): >= 7 days after the last dose of agent; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Corticosteroids: if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell Infusions (with or without total body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: >= 84 days after infusion and no evidence of graft versus host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: >= 42 days
  * Cellular therapy: >= 42 days after the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * Radiation therapy (XRT)/external beam irradiation including protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial brain metastases (BM) radiation
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131I-metaiodobenzylguanidine [MIBG]): >= 42 days after systemically administered radiopharmaceutical therapy
  * Patients must not have received prior exposure to pevonedistat; patients with prior exposure to irinotecan or temozolomide are eligible
* For patients with solid tumors without known bone marrow involvement:

  * Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
  * Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
  * Hemoglobin >= 8 g/dL
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions); these patients will not be evaluable for hematologic toxicity; at least 5 of every cohort of 6 patients on Part A1 must be evaluable for hematologic toxicity for the dose-escalation part of the study; if dose-limiting hematologic toxicity is observed, all subsequent patients enrolled must be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * Age: 6 months to < 1 years maximum serum creatinine (mg/dL): male: 0.5; female: 0.5
  * Age: 1 to < 2 years maximum serum creatinine (mg/dL): male: 0.6; female: 0.6
  * Age: 2 to < 6 years maximum serum creatinine (mg/dL): male: 0.8; female: 0.8
  * Age: 6 to < 10 years maximum serum creatinine (mg/dL): male: 1; female: 1
  * Age: 10 to < 13 years maximum serum creatinine: (mg/dL): male: 1.2; female: 1.2
  * Age: 13 to < 16 years maximum serum creatinine: (mg/dL): male: 1.5; female: 1.4
  * Age: >= 16 years maximum serum creatinine: (mg/dL) male: 1.7; female: 1.4
* Bilirubin (sum of conjugated + unconjugated) =< upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransaminase [ALT]) =< 135 U/L; for the purpose of this study, the ULN for SGPT is 45 U/L
* Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase) [AST]); =< 150 U/L; for the purpose of this study, the ULN for SGOT is 50 U/L
* Serum albumin >= 2.7 g/dL
* Shortening fraction of >= 27% by echocardiogram, or
* Ejection fraction of >= 50% by gated radionuclide study
* No supraventricular arrhythmia on electrocardiogram (EKG)
* Prolonged rate corrected QT (QTc) interval < 500 msec
* Pulse oximetry > 94% on room air if there is clinical indication for determination (e.g. dyspnea at rest)
* Patients with seizure disorder may be enrolled if on non-enzyme inducing anti-convulsants and well controlled
* Nervous system disorders (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0) resulting from prior therapy must be =< grade 2, with the exception of decreased tendon reflex (DTR); any grade of DTR is eligible
* International normalized ratio (INR) =< 1.5
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study because there is not yet available information regarding human fetal or teratogenic toxicities; pregnancy tests must be obtained in girls who are post-menarchal
* Males or females of reproductive potential may not participate unless they have agreed to practice 1 highly effective and 1 additional effective (barrier) method of contraception at the same time during the entire study treatment period and through 4 months after the last dose of study drug, or agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject; periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception
* Patients with uncontrolled high blood pressure (i.e., systolic/diastolic blood pressure > 99th percentile) are not eligible
* Patients with known cardiopulmonary disease are not eligible; cardiopulmonary disease is defined as:

  * Cardiomyopathy other than chemotherapy related changes in cardiac function that meet the eligibility requirements
  * Clinically significant arrhythmia:

    * History of polymorphic ventricular fibrillation or torsade de pointes,
    * Permanent atrial fibrillation (a fib), defined as continuous a fib for >= 6 months,
    * Persistent a fib, defined as sustained a fib lasting > 7 days and/or requiring cardioversion in the 4 weeks before screening,
    * Grade 3 a fib defined as symptomatic and incompletely controlled medically, or controlled with device (e.g. pacemaker), or ablation and
    * Patients with paroxysmal a fib or < grade (Gr) 3 a fib for period of at least 6 months are permitted to enroll provided that their rate is controlled on a stable regimen
  * Implantable cardioverter defibrillator;
  * Moderate to severe aortic and/or mitral stenosis or other valvulopathy (ongoing);
  * Pulmonary hypertension
  * Congestive heart failure class III or IV
* Patients with known hepatic cirrhosis or severe pre-existing hepatic impairment are not eligible
* Patients with uncontrolled coagulopathy or bleeding disorder are not eligible
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible; if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients must not have received enzyme-inducing anticonvulsants for at least 7 days prior to enrollment
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients who are receiving any investigational agent other than pevonedistat, including but not limited to androgens, supraphysiologic doses of corticosteroids, erythropoietin, eltrombopag, or romiplostim
* Patients who have received drugs that are strong inducers of CYP3A4 within 14 days prior to study enrollment are not eligible; while on study, concomitant use of strong CYP3A4 inhibitors, BCRP inhibitors (cyclosporine, eltrombopag, gefitinib), and UGT1A1 inhibitors, (diclofenac, ketoconazole, probenecid, silibinin, nilotinib and atazanavir) should be avoided because of potential for increased irinotecan toxicity
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients with known human immunodeficiency virus (HIV) seropositive are not eligible
* Patients with known hepatitis B surface antigen seropositive or known or suspected active hepatitis C infection are not eligible; NOTE: patients who have isolated positive hepatitis B core antibody (i.e., in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load; patients who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load
* History of allergic reactions attributed to compounds of similar chemical or biologic composition as the study agents
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer H Foster, Principal Investigator — Pediatric Early Phase Clinical Trial Network
Locations (20):
- United States (20):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A Dose Level 1: 15 mg/m^2; Part A Dose Level 2: 20 mg/m^2; Part A Dose Level 3: 25 mg/m^2; Part A Dose Level 4: 35 mg/m^2; Part A PK Dose Level 4: 35 mg/m^2: Patients with recurrent or refractory solid tumors, including CNS tumors and lymphoma, receive pevonedistat IV over 60 minutes on days 1, 8, 10, and 12, temozolomide PO daily on days 8-12, and irinotecan IV over 90 minutes on days 8-12 of cycle 1. Beginning cycle 2, patients receive pevonedistat IV over 60 minutes on days 1, 3, and 5, temozolomide PO daily on days 1-5, and irinotecan IV over 90 minutes on days 1-5. Treatment repeats every 28 days for cycle 1 and 21 days for subsequent cycles for up to 17 cycles in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Part A Dose Level 1: 15 mg/m^2 | Part A Dose Level 2: 20 mg/m^2 | Part A Dose Level 3: 25 mg/m^2 | Part A Dose Level 4: 35 mg/m^2 | Part A PK Dose Level 4: 35 mg/m^2
Started | 6 | 6 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 6 | 6 | 6
Not completed — Lack of Efficacy | 5 | 5 | 6 | 5 | 5
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A Dose Level 1: 15 mg/m^2 | Part A Dose Level 2: 20 mg/m^2 | Part A Dose Level 3: 25 mg/m^2 | Part A Dose Level 4: 35 mg/m^2 | Part A PK Dose Level 4: 35 mg/m^2 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 4 | 6 | 6 | 28
  Between 18 and 65 years | 0 | 0 | 2 | 0 | 0 | 2
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 14.5 [6 to 18] | 12 [1 to 17] | 11 [2 to 21] | 7 [5 to 15] | 16.5 [4 to 18] | 13 [1 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 4 | 1 | 3 | 11
  Male | 5 | 4 | 2 | 5 | 3 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 2 | 2 | 5
  Not Hispanic or Latino | 5 | 6 | 5 | 4 | 4 | 24
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 0 | 3 | 6
  White | 5 | 3 | 3 | 5 | 2 | 18
  More than one race | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 0 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: MTD/RP2D of Pevonedistat in Combination With Irinotecan and Temozolomide
Description: The maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) will be the maximum dose at which fewer than one-third of patients experience dose limiting toxicities.
Time Frame: Up to 28 days
Population: All Part A patients
Measure: Number; unit: mg/m^2
Groups:
- Treatment (Pevonedistat, Temozolomide, Irinotecan): Patients with recurrent or refractory solid tumors, including CNS tumors and lymphoma, receive pevonedistat IV over 60 minutes on days 1, 8, 10, and 12, temozolomide PO daily on days 8-12, and irinotecan IV over 90 minutes on days 8-12 of cycle 1.
Arm/Group | Treatment (Pevonedistat, Temozolomide, Irinotecan)
Number analyzed (Participants) | 30
mg/m^2 | 35

2. Primary Outcome: Number of Participants With Grade 3 or Greater Toxicities Associated With Pevonedistat in Combination With Irinotecan and Temozolomide
Description: Frequency of patients who experience at least one grade 3 or higher toxicity that is at least possibly attributable to pevonedistat using the Common Terminology Criteria for Adverse Events version 5.0 by dose level stratified by study part and dose level.
Time Frame: Up to 3 years 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Dose Level 1: 15 mg/m^2 | Part A Dose Level 2: 20 mg/m^2 | Part A Dose Level 3: 25 mg/m^2 | Part A Dose Level 4: 35 mg/m^2 | Part A PK Dose Level 4: 35 mg/m^2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Participants | 5 | 4 | 6 | 2 | 4

3. Primary Outcome: Half-life of Pevonedistat in Combination With Irinotecan and Temozolomide
Description: Median (Range) for the time required for the serum concentration to fall to 50% of its starting dose by dose level stratified by study part and dose level.
Time Frame: Up to 10 days
Population: All eligible patients with data collected
Measure: Median (Full Range); unit: hours
Arm/Group | Part A Dose Level 1: 15 mg/m^2 | Part A Dose Level 2: 20 mg/m^2 | Part A Dose Level 3: 25 mg/m^2 | Part A Dose Level 4: 35 mg/m^2 | Part A PK Dose Level 4: 35 mg/m^2
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
hours | 5.3 [4.7 to 7.4] | 5 [4.1 to 6.0] | 5.2 [4.0 to 5.5] | 4.7 [4.0 to 6.7] | 6.1 [3.9 to 7.9]

4. Primary Outcome: T Max of Pevonedistat in Combination With Irinotecan and Temozolomide
Description: Median (Range) for the time at which the maximum (peak) serum concentration occurs by dose level stratified by study part and dose level.
Time Frame: Up to 10 days
Population: All eligible patients with data collected
Measure: Median (Full Range); unit: hours
Arm/Group | Part A Dose Level 1: 15 mg/m^2 | Part A Dose Level 2: 20 mg/m^2 | Part A Dose Level 3: 25 mg/m^2 | Part A Dose Level 4: 35 mg/m^2 | Part A PK Dose Level 4: 35 mg/m^2
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
hours | 1. [1.0 to 1.6] | 1 [1.0 to 2.5] | 1 [0.9 to 1.4] | 1.1 [1.0 to 1.1] | 1.1 [1.0 to 1.5]

5. Primary Outcome: C Max of Pevonedistat in Combination With Irinotecan and Temozolomide
Description: Median (Range) for the maximum (peak) serum concentration by dose level stratified by study part and dose level.
Time Frame: Up to 10 days
Population: All eligible patients with data collected
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Part A Dose Level 1: 15 mg/m^2 | Part A Dose Level 2: 20 mg/m^2 | Part A Dose Level 3: 25 mg/m^2 | Part A Dose Level 4: 35 mg/m^2 | Part A PK Dose Level 4: 35 mg/m^2
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
ng/mL | 156 [87.9 to 208.0] | 218.5 [170.5 to 335.0] | 303.5 [174.0 to 365.5] | 419 [238.0 to 689.0] | 363.8 [214.0 to 2367.0]

6. Primary Outcome: AUC of Pevonedistat in Combination With Irinotecan and Temozolomide
Description: Median (range) of the area under the drug concentration over time (pre-dose and then 0, 1, 2, 4, 6-8, and 24-hours post-dose infusion) curve stratified by study part and dose level.
Time Frame: Up to 10 days
Population: All eligible patients with data collected
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Part A Dose Level 1: 15 mg/m^2 | Part A Dose Level 2: 20 mg/m^2 | Part A Dose Level 3: 25 mg/m^2 | Part A Dose Level 4: 35 mg/m^2 | Part A PK Dose Level 4: 35 mg/m^2
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
hr*ng/mL | 803 [608.0 to 1010.0] | 973.5 [865.0 to 1928.0] | 1340 [990.0 to 1890.0] | 2018.5 [1505.0 to 2535.0] | 1957 [1583.0 to 5733.0]

7. Primary Outcome: Clearance of Pevonedistat in Combination With Irinotecan and Temozolomide
Description: Median (Range) for the rate of elimination of the drug by dose level stratified by study part and dose level.
Time Frame: Up to 10 days
Population: All eligible patients with data collected
Measure: Median (Full Range); unit: L/hr/m^2
Arm/Group | Part A Dose Level 1: 15 mg/m^2 | Part A Dose Level 2: 20 mg/m^2 | Part A Dose Level 3: 25 mg/m^2 | Part A Dose Level 4: 35 mg/m^2 | Part A PK Dose Level 4: 35 mg/m^2
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
L/hr/m^2 | 18.8 [14.8 to 24.7] | 20.8 [10.6 to 23.3] | 18.9 [13.2 to 25.4] | 17.5 [13.8 to 23.3] | 17.9 [10.2 to 22.1]

8. Secondary Outcome: Anti-tumor Activity of Pevonedistat in Combination With Irinotecan and Temozolomide
Description: Frequency of disease response (best overall response of partial or complete response) assessed per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR by dose level.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Dose Level 1: 15 mg/m^2 | Part A Dose Level 2: 20 mg/m^2 | Part A Dose Level 3: 25 mg/m^2 | Part A Dose Level 4: 35 mg/m^2 | Part A PK Dose Level 4: 35 mg/m^2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Participants | 1 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Part A Dose Level 1: 15 mg/m^2 | Part A Dose Level 2: 20 mg/m^2 | Part A Dose Level 3: 25 mg/m^2 | Part A Dose Level 4: 35 mg/m^2 | Part A PK Dose Level 4: 35 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 5/6 | 4/6 | 6/6 | 2/6 | 4/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Dose Level 1: 15 mg/m^2 (N=6) | Part A Dose Level 2: 20 mg/m^2 (N=6) | Part A Dose Level 3: 25 mg/m^2 (N=6) | Part A Dose Level 4: 35 mg/m^2 (N=6) | Part A PK Dose Level 4: 35 mg/m^2 (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Fever (General disorders) | 0 | 0 | 1 | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 0 | 1 | 0
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Ileal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 5 | 0 | 2 | 1 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 3 | 1 | 2 | 2 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Premature menopause (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Surgical and medical procedures - Other, tumor resection surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
White blood cell decreased (Investigations) | 5 | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Dose Level 1: 15 mg/m^2 (N=6) | Part A Dose Level 2: 20 mg/m^2 (N=6) | Part A Dose Level 3: 25 mg/m^2 (N=6) | Part A Dose Level 4: 35 mg/m^2 (N=6) | Part A PK Dose Level 4: 35 mg/m^2 (N=6)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 3 | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 4 | 5 | 5 | 4 | 3
Alkaline phosphatase increased (Investigations) | 3 | 1 | 0 | 1 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 4 | 2
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 6 | 4 | 6 | 6 | 5
Anorexia (Metabolism and nutrition disorders) | 3 | 4 | 3 | 3 | 3
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 6 | 5 | 2 | 4
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 1 | 2
Blood and lymphatic system disorders - Other, RBC DECREASED (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 2
Blurred vision (Eye disorders) | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
CPK increased (Investigations) | 0 | 0 | 1 | 0 | 0
Cardiac disorders - Other, (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Cholesterol high (Investigations) | 0 | 0 | 1 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 3 | 3 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1 | 1
Creatinine increased (Investigations) | 2 | 0 | 1 | 1 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 1 | 1 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 4 | 6 | 3 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2
Ear and labyrinth disorders - Other, (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Edema limbs (General disorders) | 0 | 1 | 0 | 1 | 2
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Eye disorders - Other, DIPLOPIA (Eye disorders) | 1 | 0 | 0 | 0 | 0
Eye disorders - Other, PTOSIS (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eyelid function disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0
Facial muscle weakness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 3 | 2 | 3 | 5
Fecal incontinence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Fever (General disorders) | 2 | 2 | 3 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 0 | 1 | 0
GGT increased (Investigations) | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 2 | 1 | 2 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal disorders - Other, HYPERSALIVATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal disorders - Other, TONGUE ITCHINESS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Growth hormone abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 3 | 1 | 2
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 1 | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Hemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hot flashes (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 4 | 4 | 3 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 2 | 2 | 1 | 3
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 2 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 0 | 4 | 2 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2 | 2 | 4 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 2 | 3 | 2 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 4 | 4 | 3 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 2 | 3 | 2 | 1
Hypotension (Vascular disorders) | 3 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 2 | 2 | 0 | 0
Infections and infestations - Other, THRUSH (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infections and infestations - Other, c. diff infections (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infusion related reaction (General disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1
Investigations - Other, (Investigations) | 0 | 0 | 0 | 0 | 1
Investigations - Other, BICARBONATE SERUM LOW (Investigations) | 0 | 1 | 0 | 0 | 0
Investigations - Other, Blood Bicarbonate Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Investigations - Other, Decreased chloride (Investigations) | 0 | 0 | 1 | 0 | 0
Investigations - Other, ELEVATED BUN (Investigations) | 0 | 1 | 0 | 0 | 0
Investigations - Other, ELEVATED LDH (Investigations) | 0 | 1 | 0 | 0 | 0
Investigations - Other, LDH increased (Investigations) | 0 | 0 | 1 | 0 | 0
Investigations - Other, LOW BICARBONATE (Investigations) | 0 | 1 | 0 | 0 | 0
Investigations - Other, Low CO2 (Investigations) | 0 | 0 | 1 | 0 | 0
Investigations - Other, Low Chloride (Investigations) | 0 | 0 | 1 | 0 | 0
Investigations - Other, PT elevated (Investigations) | 0 | 0 | 1 | 0 | 0
Iron overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
Keratitis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Localized edema (General disorders) | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lymphedema (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 4 | 3 | 3 | 4 | 3
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Metabolism and nutrition disorders - Other, Chloride Increased (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Metabolism and nutrition disorders - Other, vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Movements involuntary (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Muscle weakness left-sided (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle weakness right-sided (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Musculoskeletal and connective tissue disorder - Other, AXIAL SKELETAL INVOLVEMENT WITH MULTIPLE BON (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, RIB CAGE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, SCAPULA PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, SKULL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 5 | 4 | 3 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Nervous system disorders - Other, (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Nervous system disorders - Other, Cholinergic reaction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Nervous system disorders - Other, HYPERALGESIA (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Nervous system disorders - Other, Intermittent facial numbness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 4 | 4 | 3 | 4 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Oculomotor nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 3 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1
Papulopustular rash (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 2
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 3 | 4 | 4 | 1 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Precocious puberty (Endocrine disorders) | 0 | 1 | 1 | 0 | 0
Premature menopause (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Psychiatric disorders - Other, (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Psychiatric disorders - Other, DELIBERATE SELF-CUTTING (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary valve disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Renal and urinary disorders - Other, DYSURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Reproductive system and breast disorders - Other, vaginal odor (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, TACHYPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rhinitis infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 2 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 1 | 4 | 2 | 0
Skin and subcutaneous tissue disorders - Other, SCARRING (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Spasticity (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Surgical and medical procedures - Other, Portacath placement (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Tricuspid valve disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2 | 1
Unequal limb length (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1
Vaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Vascular disorders - Other, (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 4 | 4 | 2 | 5
Weight gain (Investigations) | 1 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 0 | 0 | 1 | 0 | 1
White blood cell decreased (Investigations) | 5 | 6 | 5 | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT03323034/Prot_SAP_000.pdf